CLINICAL TRIAL: NCT02369913
Title: A Metabolomic Approach to Probing Myocardial Fuel Shifts in Human Heart Failure
Status: Withdrawn | Type: Observational
Why Stopped: The Study has been officially closed with the IRB
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 201401007
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Heart failure subjects: Heart failure subjects undergoing cardiac resynchronization will have a blood drawn for this study.
  Interventions: Other: Blood Drawn
- Heart arrhythmia patients: Heart arrhythmia patients undergoing ablation will have a blood drawn for this study.
  Interventions: Other: Blood Drawn

INTERVENTIONS:
Other: Blood Drawn — Both groups will have 1 teaspoon of blood drawn for analysis.

SUMMARY:
This proposal is designed to test the hypothesis that humans shift to reliance on ketone bodies as a cardiac fuel source during the development of HF. The investigator also propose that this shift to ketone utilization can be detected by metabolomic profiling of blood.

Specific Aim 1: To determine if the failing human heart exhibits increased extraction of blood-borne ketone bodies. Ketone bodies will be measured in coronary sinus, arterial, and central venous blood samples to determine AV differences. The HF group will be comprised of patients undergoing cardiac resynchronization therapy with an implantable cardioverter-defibrillator. The Control group will be compromised of patients without evidence of structural heart disease who are undergoing catheter ablation for supraventricular tachycardia.

Specific Aim 2: To determine whether blood samples from humans with HF display metabolomic signatures indicative of increased myocardial ketone body utilization. Quantitative targeted metabolomics will be performed on the samples described in Aim 1 to determine if metabolite markers (e.g. C4-OH acylcarnitine, acetylcarnitine, succinate) found to be associated with increased myocardial ketone body oxidation in animal models are increased in the human HF group compared to the controls.

DETAILED DESCRIPTION:
After subjects agree to participate in this study and are scheduled to have cardiac resynchronization therapy, the research personnel will take 1 teaspoon of blood before and after the scheduled cardiac procedure for comparison.

Once subjects agree to participate in this study and are scheduled to have a catheter ablation procedure, research personnel will take 1 teaspoon of blood during the scheduled cardiac procedure.

These samples will be taken from catheters already placed during the scheduled cardiac procedure.

Blood will be sent to a lab at the Sanford-Burnham Metabolomics Core Facility in Orlando, Florida for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiac resynchronization therapy
* Undergoing sinus cannulation

Exclusion Criteria:

* NYHA class II-IV heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing cardiac resynchronization therapy or receiving a catheter ablation procedure.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Increased extraction of blood-borne ketone bodies | 1 day
  Ketone bodies will be measured in coronary sinus, arterial, and central venous blood samples to determine AV differences
Determine whether heart failure blood samples display metabolomic signatures | 1 day
  Quantitative targeted metabolomics will be performed on the samples described in Outcome 1 to determine if metabolite markers (e.g. C4-OH acylcarnitine, acetylcarnitine, succinate) found to be associated with increased myocardial ketone body oxidation in animal models are increased in the human HF group compared to the controls.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Handberg, PhD, Principal Investigator — University of Florida
Locations (1):
- University of florida, Gainesville, Florida, United States